CLINICAL TRIAL: NCT01558466
Title: Early Combined Use of Inhaled Nitric Oxide and Oral Sildenafil on the Outcome of Pulmonary Hypertension in New Born Infants
Brief Title: Sildenofil in Persistent Pulmonary Hypertension in Newborns
Acronym: Sildeno
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10228/10
Record Dates: First submitted 2012-03-11; First posted 2012-03-20 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Persistent Fetal Circulation Syndrome
Keywords: newborn; INO; Sildenafil; PPHN
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome | interventions — Sildenafil Citrate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A - Placebo (Placebo Comparator): iNO combined with placebo will be administered
  Interventions: Drug: diluent
- Group B- Sildenafil (Active Comparator): iNO combined with Sildenafil
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — 50 mg tablet will be thoroughly crushed into powder form and diluted in 10 ml ora base suspension syrup agent and a dilution will be performed to prepare 5 mg/ml. All doses required for 48 hours will be available; solutions will be stored at 2-8 degrees C where solution should be stable for at least a month.
  Other Names: Viagra
  Arms: Group B- Sildenafil
Drug: diluent — The placebo will have an equal volume of diluent - Orabase syrup of the same colour and viscosity as the active comparator. Infants in this group will receive normal saline as placebo every 6 hours
  Other Names: Normal saline
  Arms: Group A - Placebo

SUMMARY:
This study hopes to evaluate the effectiveness of early combined use of Sildenafil and nitric oxide (iNO) in newborns with Persistent pulmonary hypertension (PPHN) and or hypoxemic respiratory failure and assess whether this would improve oxygenation, improve time on mechanical ventilation for these babies and also prevent rebound hypoxic episodes.

DETAILED DESCRIPTION:
PPHN is characterized by hyper reactivity of the muscle layer in pulmonary arterioles and right to left shunt across the ductus arteriosus and the foramen ovale in the absence of structural heart defects. It could also include right ventricle dysfunction in many cases. The reported incidence of this disease is 0.43 to 6.8/1000 live new born infants with a mortality of 10-20%.

The main objective of therapy in PPHN is to reduce pulmonary vascular resistance. To this purpose, inhaled nitric oxide has been used in developed and several under developed countries. However 30-40% of these patients do not respond to this therapy. Extra corporeal membrane oxygenation is also useful but is an invasive therapy in PPHN with serious adverse effects reported. Recently Sildenafil has been evaluated as an alternative or adjunctive pulmonary vasodilator. It inhibits phosphodiesterase type 5 and elevates the concentration of cyclic guanosine monophosphate in the muscle cells of pulmonary vessels, which in turn decreases pulmonary vascular resistance.

The FDA in the USA has recently approved the use of Sildenafil for use in adults with PPHN.

Recently 3 clinical trials have evaluated Sildenafil versus Placebo or control in newborns with PPHN,all of them showing a significant improvement in oxygenation index, decreased mortality and reduced risk of rebounds after discontinuing iNO. The use of Sildenafil in treating PPHN secondary to Chronic lung disease in older infants had been receiving significant attention over the last few years.

At HMC, Women's hospital, the number of deliveries average 15,000 to 16,000 per year with an admission rate to the NICU of about 10%. The number of PPHN cases admitted to our NICU ranges between 14-20 cases per year.

In this study the investigators plan to compare the effectiveness of the use of early combined Sildenafil and iNO in newborns with PPHN and or hypoxemic respiratory failure and whether it would improve oxygenation, decrease the time spent in mechanical ventilation and prevent rebound hypoxic episodes.

ELIGIBILITY:
Inclusion Criteria:

1. Newborn infants of post natal age less than 48 hours
2. Gestational age equal to or more than 34 weeks
3. Oxygen index of more than or equal to 20 (moderately ill infants)
4. Radiological, clinical and biochemical evidence of acute hypoxic respiratory failure
5. Surfactant therapy has been established when indicated
6. Presence of arterial line

Exclusion Criteria:

1. Congenital diaphragmatic hernia
2. Major congenital abnormalities
3. Significant congenital heart disease
4. Cyanotic congenital heart disease

Ages: 36 Weeks to 41 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-11 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Oxygen index | 7 days after birth and admission to the NICU
  OI= PaO2 X FiO2/100( Absolute values and change from baseline measurement after first dose, measured every 6 hours for 7 days while on therapy. Improvement in OI is defined as decrease in OI of 20% from the previously calculated value.
A-a gradient | 7 days after admission to the NICU
  Alveolar arterial oxygen difference gradient
Hemodynamic parameters | 7 days
  Hemodynamic parameters ( absolute values and change from baseline measured after the first dose, after 24 hours, after 36 hours, and after 48 hours and every 12 hours thereafter for a total of 7 days while receiving therapy and 7 days after the end of treatment including :
  1. Heart rate, mean blood pressure, respiratory rate, oxygen saturation and blood gas b. Pulmonary arterial pressure in mm Hg measured by echocardiography c. cArdiac output in liter/kg/min d. Oxygenation ( PaO2) and FiO2 requirement

SECONDARY OUTCOMES:
Days of hospitalization | 7 days after admission to the NICU
  Length of hospitalization and mortality, morbidity, ventialtion dats , adverse events
mortality | 28 days of life
  All cause mortality within 28 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Husam Salama, MD, Principal Investigator — Hamad Medical Corporation, Doha, Qatar
Locations (1):
- Women's hospital, NICU, Doha, Qatar, Qatar